CLINICAL TRIAL: NCT03061864
Title: The Periviable Birth Plan: A Randomized Control Trial Evaluating an Intervention to Decrease Maternal Anxiety and Stress
Brief Title: The Periviable Birth Plan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Paul Burcher Md, PhD, Principal Investigator, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4622
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy, High Risk; Parturition Complication as Antepartum Condition; Anxiety; PTSD; PreTerm Birth
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Counseling (No Intervention): Patients at risk of delivery between 20 and 25+6 weeks gestation will receive the normal counseling from Ob/gyn and Neonatology.
- Periviable Birth Plan (Experimental): Patients at risk of delivery between 20 and 25+6 weeks gestation will receive the normal counseling from Ob/gyn and Neonatology with completion of the written periviable birth plan.
  Interventions: Behavioral: Periviable Birth Plan

INTERVENTIONS:
Behavioral: Periviable Birth Plan
  Arms: Periviable Birth Plan

SUMMARY:
Pregnant women who are at risk of delivering their infants in the periviable period can suffer a large amount of stress and anxiety. Moreover, many women feel a loss of control over their own pregnancy. There is some evidence that more counseling and planning can help reduce maternal stress and anxiety. Patients at risk of delivering in the periviable period will be randomized to either receive standard counselling or to complete the periviable birth plan.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old.
* Currently Pregnant
* High risk of pre-term birth in the periviable period 20+0 to 25+6 wga

Exclusion Criteria:

* Intrauterine Fetal Demise (prior to admission)
* Inability to read or communicate in english

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08

PRIMARY OUTCOMES:
Change in Anxiety Scores | Time of Delivery and One Year
  Patients will complete State Trait Anxiety Inventory questionnaire at the time of delivery and again at 1 year from completion of the first questionnaire. Those that do not deliver in the periviable period will complete the first questionnaire at 27 weeks gestation.
Change in PTSD Scores | Time of Delivery and One Year
  Patients will complete Impact of Events Scale questionnaire at the time of delivery and again at 1 year from completion of the first questionnaire. Those that do not deliver in the periviable period will complete the first questionnaire at 27 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Burcher, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No